CLINICAL TRIAL: NCT04156789
Title: Obstructive Sleep Apnoea in Sarcoidosis: A Cross-sectional Observational Study
Brief Title: Obstructive Sleep Apnoea in Sarcoidosis
Acronym: OSASA
Status: Completed | Type: Observational
Sponsor: Malcolm Kohler (Other)
Responsible Party: Sponsor-Investigator, Malcolm Kohler, Head of the department of pulmonology, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2019-01604
Record Dates: First submitted 2019-10-30; First posted 2019-11-08 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Sarcoidosis; Obstructive Sleep Apnea; Fatigue; Sleepiness
MeSH Terms: conditions — Sarcoidosis; Sleep Apnea, Obstructive; Fatigue; Sleepiness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling to assess inflammation marker: sIL-2-Receptor, Neopterin, Angiotensin Converting Enzyme (ACE) and hsCRP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcoidosis group: Subjects with a definite diagnosis of sarcoidosis according to international ATS and WASOG guideline
  Interventions: Diagnostic Test: Home sleep apnea testing
- Control group: Control subjects have no sarcoidosis and will be sex, age (± 3 years), height (± 20 cm), and weight (± 15 kg) matched to sarcoidosis patients.
  Interventions: Diagnostic Test: Home sleep apnea testing

INTERVENTIONS:
Diagnostic Test: Home sleep apnea testing — Sarcoidosis patients and control subjects will undergo one night of home sleep apnea testing using ApnoeaLinkTM Plus device (ResMed Corporation, Poway, Calif). The device records the patient's nasal respiratory pressure signal as a surrogate of nasal flow, respiratory movements by a thoracic impedance belt, and finger pulse oximetry. The results of the sleep study will be scored automatically with dedicated software (ResMed Corporation, Poway, Calif), and manually reviewed to ensure data accuracy.

SUMMARY:
Sarcoidosis is a multisystemic granulomatous disease of unknown origin. Fatigue is a common problem in sarcoidosis affecting between 50% and 80% of patients, and thus represents a major impairment of their quality of life.

The findings of recent studies suggest a high prevalence of obstructive sleep apnoea (OSA) in patients with sarcoidosis, estimating a range from 17% to 67%. Pathomechanisms leading to this increased OSA prevalence are still unclear, yet likely to be multifactorial including sarcoid myopathy and neuropathy leading to impaired integrity of the upper airways as well as corticosteroid induced obesity.

While both diseases, Sarcoidosis and OSA, could lead to fatigue and excessive daytime sleepiness (EDS) the current managing strategies differ significantly. OSA patients are mostly treated with continuous positive airway pressure (CPAP) whereas sarcoidosis associated fatigue may require increased immunosuppressive therapy. Little is known about treatment of fatigue and sleepiness in patients suffering from both conditions.This study aims to close this knowledge gap and define prevalence of OSA in a swiss cohort with sarcoidosis patients.

Therefore, we plan a prospective, observational, controlled study to investigate the prevalence of sleepiness, fatigue, life quality and obstructive sleep apnoea in patients with Sarcoidosis.

Patients treated in the University Hospital Zurich due to sarcoidosis will be invited by letter to take part in this study. After confirmed consent and baseline assessments at the University Hospital Zurich, these patients will undergo a single night, in-home sleep study to assess possible OSA.

Sleepiness and fatigue specific questionnaires and in-home respiratory polygraphy (oRP) are obtained in all subjects. To assess inflammation status and other conditions connected to sleepiness like hypothyroidism and anaemia, sarcoidosis patients will undergo blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Sarcoidosis group: Subjects with a definite diagnosis of sarcoidosis according to international ATS and WASOG guideline.
* Informed consent
* 18 years or above
* Control group: No sarcoidosis, no OSA

Exclusion Criteria:

* Moribund or severe disease prohibiting protocol adherence
* Continuous positive airway pressure treatment for OSA at baseline
* Use of oxygen therapy or home ventilation
* Physical or intellectual impairment precluding informed consent or protocol adherence
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sarcoidosis group: Subjects with a definite diagnosis of sarcoidosis according to international ATS and WASOG guideline
  vs
  Control group: matched control subjects without sarcoidosis
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of OSA in sarcoidosis patients compared to matched controls | through one sleep study night
  Conventional thresholds according to the American Academy of Sleep Medicine Task Force of AHI ≥5, ≥15 and ≥30 will be used to define mild, moderate and severe OSA respectively. OSA prevalence will be compared between both groups.

SECONDARY OUTCOMES:
Apnoea-Hypopnea Index (AHI) | through one sleep study night
  AHI will be compared between both groups.
Fatigue Severity Scale (FAS) | one day
  FAS will be compared between both groups. Score ranges from 10 to 50 points with 50 points presenting the most severe form of fatigue.
Blood pressure | one day
  Blood pressure will be compared between both groups.
Lung function test | one day
  Lung function tests will be compared between both groups.
Puls wave analysis | one day
  Applanation-derived augmentation index (AIx) will be compared between both groups.
Interleukin-2 blood levels | one day
  Association between Interleukin-2 blood levels and OSA severity (AHI) and excessive daytime sleepiness (ESS) in sarcoidosis will be assessed.
Oxygen-Desaturation Index (ODI) | through one sleep study night
  ODI will be compared between both groups.
Epworth Sleepiness Scale (ESS) | one day
  ESS will be compared between both groups. The test measures subjective sleepiness. The scale ranges from 0 to 24 points. More points indicate higher sleepiness.
Functional outcomes of sleep questionnaire (FOSQ) | one day
  FOSQ will be compared between both groups. The score ranges from 5 to 20 points. Higher scores indicate better functional status.
Short-form-36 (SF-36) | one day
  SF-36 will be compared between both groups. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Patient Health Questionnaire (PHQ) Module 9 | one day
  PHQ 9 will be compared between both groups. The test results range between 0 and 27 points. Higher scores indicate severe forms of depression.
NoSAS-Score | one day
  NoSAS-Score will be compared between both groups. The score ranges from 0-17 points. The patient has a high probability of sleep disordered breathing if he has a NoSAS-Score of 8 or higher.
Heart rate | one day
  Heart rate will be compared between both groups
Neopterin blood level | one day
  Association between Neopterin blood levels and OSA severity (AHI) and excessive daytime sleepiness (ESS) in sarcoidosis will be assessed.
C-reactive protein (CRP) blood levels | one day
  Association between CRP blood levels and OSA severity (AHI) and excessive daytime sleepiness (ESS) in sarcoidosis will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, Prof, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Roeder M, Sievi NA, Schneider A, Osswald M, Malesevic S, Kolios A, Nilsson J, Kohler M, Franzen D. The prevalence of obstructive sleep apnea in sarcoidosis and its impact on sleepiness, fatigue, and sleep-associated quality of life: a cross-sectional study with matched controls (the OSASA study). J Clin Sleep Med. 2022 Oct 1;18(10):2415-2422. doi: 10.5664/jcsm.10140. PMID 35855534